CLINICAL TRIAL: NCT06975930
Title: Outcomes of Different Techniques of Aortoostial Coronary Intervention Assessed by Coronary Computed Tomography Angiography
Acronym: Aortoostial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdalla Aly, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Aorto-ostial coronary PCI
Record Dates: First submitted 2025-04-27; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Coronary Interventions
Keywords: coronary interventions
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): patients who will undergo 2D convnetional angiography Aorto-ostial coronary stenting
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)
- Floating Wire group (Active Comparator): Patients who will undergo Aorto-ostial coronary stenting with Floating wire technique
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — Patients with Aortoostial coronary lesion undergoing PCI will be blindly randomized into 2 groups Conventional group: patients who will undergo 2D convnetional angiography Aorto-ostial coronary stenting.
  Floating Wire group: Patients who will undergo Aorto-ostial coronary stenting with Floating wire technique.
  Other Names: PCI

SUMMARY:
Aorto-ostial coronary lesions (AOL) are defined as a stenosis >50% within 3 mm of the orifice of the right coronary artery (RCA) or left main coronary artery (LMCA).

The prevalence of AOL varies according to the studied population and is more common in the RCA.

Aorto-ostial lesions commonly have a unique three-dimensional funnel-shaped morphology with a variable angle of takeoff of the coronary artery from the aorta.

Percutaneous treatment of AOL is challenging due to a variety of factors which include unfavorable lesion histology, complex 3D anatomy, inability of conventional angiography to reliably delineate the aorto-ostial plane and guide the intervention and unsuitability of current tubular stent designs for this lesion subset.

Coronary computed tomography angiography (CCTA) clearly defines AOL anatomy, its relation to the aortic wall and the degree of plaque calcification.

CCTA is uniquely suited to assess the accuracy of AOL stent implantation. While conventional single wire technique is the most commonly used approach for AOL stenting, An approach uses an accessory free floating guide-wire placed within the aortic sinus to mark the aorto-ostial plane and prevent entry of the catheter into the coronary artery is called floating wire technique & is being used now.

Aim of work: 1-Comparison between 2D angiography versus Floating wire technique regarding aorto-ostial stent implantation site within the AOLZ assessed by CCTA .

2- Short term outcomes regading MACE in both groups including : myocardial infarction (MI), stroke, all-cause mortality and target vessel revascularisation (TVR).

* Type of the study: This is a randomized prospective cross sectional study
* Duration of the study: Patients will be recruited over a period of 12 months.
* Study Population: The study will include all patients who will undergo aorto-ostial coronary stenting & patients will be categorized into 2 groups Group A:patients who will undergo 2D convnetional angiography Aorto-ostial stenting.

Group B: Patients who will undergo Aorto-ostial stenting with Floating wire technique.

Patients will undergo CCTA to detect geographic miss within 6 months of stent impalntation.

Both groups will be followed up clinically to detect adverse clinical outcomes such as AMI, recurrent chest pain,….etc.

Methdos:

Optimal AOL stenting requires placement of the entire circumference of the proximal stent edge within the aorto-ostial landing zone (AOLZ), defined as the area along the axis of the coronary artery located within 1 mm of the aorto-ostial plane.

Stent geographic miss may be diagnosed when at least a segment of the circumference of the proximal stent edge is located proximal or distal to the AOLZ.

Accurate AOL stent implantation is crucial. If geographic miss was attributed to the angulated vessel take-off from the aorta preventing precise localisation of the cylindrical stent structure within the constraints of the AOLZ, it is defined as anatomy-dependent.

Geographic miss in which all aspects of the proximal stent edge extended beyond the AOLZ either proximally or distally was attributed to incorrect implantation of the stent and was defined as procedure-dependent.

DETAILED DESCRIPTION:
Aorto-ostial coronary lesions (AOL) are defined as a stenosis >50% within 3 mm of the orifice of the right coronary artery (RCA) or left main coronary artery (LMCA).

The prevalence of AOL varies according to the studied population and is more common in the RCA.

Aorto-ostial lesions commonly have a unique three-dimensional funnel-shaped morphology with a variable angle of takeoff of the coronary artery from the aorta.

Percutaneous treatment of AOL is challenging due to a variety of factors which include unfavorable lesion histology, complex 3D anatomy, inability of conventional angiography to reliably delineate the aorto-ostial plane and guide the intervention and unsuitability of current tubular stent designs for this lesion subset.

Coronary computed tomography angiography (CCTA) clearly defines AOL anatomy, its relation to the aortic wall and the degree of plaque calcification.

CCTA is uniquely suited to assess the accuracy of AOL stent implantation. Rubinshtein et al. recently analyzed cases of AOL stenting with CCTA. While review of the procedural angiograms suggested that stent positioning was satisfactory in 95% of the cases, CCTA revealed geographic miss in 87%. Sixty percent of the cases of geographic miss were classified as anatomy-dependent and 40% as procedure-dependent.

While conventional single wire technique is the most commonly used approach for AOL stenting, Szabo proposed a technique whereby an accessory guide-wire was passed through the most proximal stent cell and placed within the aorta, thereby preventing deep insertion of the stent into the vessel beyond the aorto-ostial plane.

Despite initial enthusiasm for this technique, it may lead to stent deformation and dislodgement.

A similar approach uses an accessory free floating guide-wire placed within the aortic sinus to mark the aorto-ostial plane and prevent entry of the catheter into the coronary artery.

Aim of work: 1-Comparison between 2D angiography versus Floating wire technique regarding aorto-ostial stent implantation site within the AOLZ assessed by CCTA .

2- Short term outcomes regading MACE in both groups including : myocardial infarction (MI), stroke, all-cause mortality and target vessel revascularisation (TVR).

* Type of the study: This is a randomized prospective cross sectional study
* Duration of the study: Patients will be recruited over a period of 12 months.
* Study Population: The study will include all patients who will undergo aorto-ostial coronary stenting & patients will be categorized into 2 groups Group A:patients who will undergo 2D convnetional angiography Aorto-ostial stenting.

Group B: Patients who will undergo Aorto-ostial stenting with Floating wire technique.

Patients will undergo CCTA to detect geographic miss within 6 months of stent impalntation.

Both groups will be followed up clinically to detect adverse clinical outcomes such as AMI, recurrent chest pain,….etc.

Methdos:

Study definitions … AOLZ defined as the area along the axis of the coronary artery located within 1 mm of the aorto-ostial plane.

Optimal AOL stenting requires placement of the entire circumference of the proximal stent edge within the aorto-ostial landing zone (AOLZ), defined as the area along the axis of the coronary artery located within 1 mm of the aorto-ostial plane.

Stent geographic miss may be diagnosed when at least a segment of the circumference of the proximal stent edge is located proximal or distal to the AOLZ.

Accurate AOL stent implantation is crucial. Proximal geographic miss with protrusion of the stent into the aorta may hinder future catheter access to the coronary artery. Distal geographic miss may leave part of the AOL uncovered by stent struts and increase the likelihood of restenosis.

If geographic miss was attributed to the angulated vessel take-off from the aorta preventing precise localisation of the cylindrical stent structure within the constraints of the AOLZ, it is defined as anatomy-dependent.

Geographic miss in which all aspects of the proximal stent edge extended beyond the AOLZ either proximally or distally was attributed to incorrect implantation of the stent and was defined as procedure-dependent.

All patients will be subjected to:

A. Full history taking B. Twelve lead ECG. C. Collecting baseline venous blood samples for Random blood glucose, serum urea & creatinine, Complete blood count, PT, PC & INR.

D. Echocardiography E. CA & PCI: All patients will be blindly randomized into the 2 groups with assessment of amount of dye needed & radiation dose.

After 3-6 months all patient will be subjected to new CA if possible specially if symptomatic for assessment of :- Significant ISR, need of further re-vasculariztion & difficulty of reengagment F. CCTA: To assess optimal stent implantation in AOLZ, partial or complete geographic miss.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old who have Aorto-ostial lesions and undergo Aorto-ostial stenting whether they have ACS or CCS.

Exclusion Criteria:

* All patients who refused CCTA or refused participation in the study.
* Patients with previous Aorto-ostial stents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Conventional Angiography vs Floating Wire technique in Aorto-ostial coronary PCI. | 6 months
  Comparison between Aorto-ostial coronary intervention (PCI) using 2D angiography versus Floating wire technique regarding aorto-ostial stent implantation site within the AOLZ which will be assessed by Coronary Computed Tomography Angiography.

SECONDARY OUTCOMES:
Short term MACE. | 6 months
  Short term outcomes regarding Major Adverse Cardiac Events in both groups including : myocardial infarction (MI), stroke, all-cause mortality and target vessel revascularization (TVR).

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University Heart Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year